CLINICAL TRIAL: NCT01547793
Title: End-Alveolar Carbon Monoxide as a Measure of Erythrocyte Survival and Hemolytic Severity in Sickle Cell Disease
Brief Title: Carbon Monoxide Levels and Sickle Cell Disease Severity
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120069; 12-H-0069
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2015-11-04

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia; Anemia, Sickle Cell
Keywords: Hemolytic Severity; Erythrocyte; Sickle Cell Disease; SD
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Some people with sickle cell disease have different health problems than others. This may be related to how easily and frequently the red blood cells break apart in the blood. Researchers want to test breath and blood samples from people with sickle cell disease to look for very small amounts of carbon monoxide, which is produced when red blood cells break apart. They will compare these results with breath samples from healthy volunteers. Studying different levels of carbon monoxide may help predict what health problems a person with sickle cell disease may get. It may also provide more information on possible treatments.

Objectives:

- To study breath carbon monoxide levels and their possible relation to the severity of sickle cell disease.

Eligibility:

* Individuals at least 18 years of age with sickle cell disease.
* Healthy volunteers who are matched for age, sex, and race with the sickle cell disease group.

Design:

* Participants will be screened with a medical history.
* Participants with sickle cell disease will provide a blood sample and have a heart function test. They will also breathe into a bag to provide an exhaled breath sample.
* Healthy volunteers will provide an exhaled breath sample.
* No treatment or care will be provided as part of this study.

DETAILED DESCRIPTION:
Sickle cell disease is an autosomal recessive disorder and the most common genetic disease affecting African-Americans. Approximately 0.15% of African-Americans are homozygous for sickle cell disease, and 8% have sickle cell trait. Hemoglobin S polymerization leads to red cell rigidity, microvascular obstruction, inflammation, and end-organ ischemic injury. Our published data indicate that up to 50% of sickle cell patients have vascular dysfunction due to impaired bioavailability of endogenous nitric oxide, due in large part to scavenging of nitric oxide by cell-free hemoglobin. In previous studies we have demonstrated that steady-state serum LDH is strongly associated with 1) other markers of intravascular hemolysis including plasma cell-free hemoglobin and arginase levels, 2) levels of soluble endothelial adhesion molecules, and 3) an impaired vasodilatory response to an NO donor. Further, significant steady-state LDH elevation identified a subset of patients in our cohort as well as the CSSCD cohort at increased risk for developing pulmonary hypertension, cutaneous leg ulceration, priapism, and early death. Previous biochemical studies have demonstrated significant transient increases in serum LDH and plasma hemoglobin levels during VOC, and this presumed hyperhemolysis has been confirmed by 51Cr labeled RBC studies that revealed further decreases in RBC survival during VOC. However, serum LDH levels are not a specific biomarker of hemolysis, and furthermore these observations on RBC survival have not been correlated with markers of intravascular hemolysis at baseline in patients with sickle cell disease in order to confirm the presence of chronic hyperhemolysis subphenotypes in sickle cell disease as posited in our previous work.

The current gold standards of random and cohort labeling of RBCs used to quantitate RBC survival suffer from many technical drawbacks that make them impractical for routine clinical use. The production rate of expired CO has previously been used to assess RBC survival, based upon the principal that virtually all CO produced in human beings results from cleavage of the ?-methene bond of heme and is completely excreted via the lungs. Because RBC destruction accounts for approximately 80% of heme turnover in the body, endogenous CO production can be used as a quantitative indicator of RBC life span. Furne et al have previously reported on the development of a simple, rapid, and noninvasive method for determining RBC life span based on measurement of exhaled alveolar CO concentration immediately upon awakening corrected for atmospheric CO, as determined with a device that simulates the body s equilibration with CO with results comparable to standard labeling techniques. We propose that this methodology could also provide a quantitative, simple, and noninvasive test to study the RBC life span and thus rate of hemolysis in those patients with sickle cell disease.

This trial will aim to 1) establish the use of end-alveolar CO concentration as a quantitative measure of RBC life span and hemolytic rate in subjects with sickle cell disease; 2) investigate the association between end-alveolar CO concentration-derived RBC life span and laboratory measures of hemolytic severity; and 3) investigate the association between end-alveolar CO concentration-derived RBC life span and the incidence of various clinical sequelae of sickle cell disease.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

All volunteer subjects must be at least 18 years of age and have provided informed, written consent for participation in this study. Eligibility in the study is determined prior to enrollment on the basis of the following inclusion and exclusion criteria. Laboratory values obtained within the preceding 60 days are sufficient for screening purposes.

INCLUSION CRITERIA for SCD Cohort

Males or females 18 years of age or older

Diagnosis of sickle cell disease (any form; electrophoretic or HPLC documentation is required)

EXCLUSION CRITERIA for SCD Cohort

Chronic scheduled transfusions

Current known pregnancy or lactation

Hemoglobin <5.0 g/dL; however, subjects may return for repeat evaluation at a later date

Currently smoking and unable to refrain from smoking for 24 hours

Subjects previously known to have conditions that may independently affect hemolytic rate:

* Infection or sepsis in the 2 weeks prior to screening
* Autoimmune hemolytic anemia
* Systemic lupus erythematosus (SLE)
* Myelodysplastic disorders, leukemia, or lymphoma
* Hereditary spherocytosis or elliptocytosis
* Severe cardiac valve dysfunction (e.g. AS, MS) or prosthetic heart valve recipients

INCLUSION CRITERIA for Controls

In order to validate the methodology for endogenous CO measurement, initially for each enrolled study subject with sickle cell disease (up to the first 30 subjects), we will recruit an African-American healthy control subject of the same gender, within 3 years of age older or younger than the matched subject with SCD. Additionally, 20 healthy control subjects will be enrolled for adenosine and any functionally or chemically related molecules blood testing, and venous blood gas testing only, to compare against subjects with sickle cell disease. Their participation in this study will consist of one blood draw of 11 mL for research laboratory testing.

EXCLUSION CRITERIA for Controls

Current pregnancy or lactation

Serum ALT values >80 IU/L

Serum creatinine >2.0 mg/dL

Hemoglobin <11.2 g/dL for females, <13.7 for males; however, subjects may return for repeat evaluation at a later date

Currently smoking

Subjects with any known form of sickle cell disease (sickle trait will NOT be excluded)

Subjects with any other known forms of hemolytic anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-01-26; Study Completion 2015-11-04

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] CROSBY WH. The metabolism of hemoglobin and bile pigment in hemolytic disease. Am J Med. 1955 Jan;18(1):112-22. doi: 10.1016/0002-9343(55)90208-4. No abstract available. PMID 13218041
- [Background] Hebbel RP. Reconstructing sickle cell disease: a data-based analysis of the "hyperhemolysis paradigm" for pulmonary hypertension from the perspective of evidence-based medicine. Am J Hematol. 2011 Feb;86(2):123-54. doi: 10.1002/ajh.21952. PMID 21264896
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Derived] van Vuren AJ, Minniti CP, Mendelsohn L, Baird JH, Kato GJ, van Beers EJ. Lactate dehydrogenase to carboxyhemoglobin ratio as a biomarker of heme release to heme processing is associated with higher tricuspid regurgitant jet velocity and early death in sickle cell disease. Am J Hematol. 2021 Sep 1;96(9):E315-E318. doi: 10.1002/ajh.26243. Epub 2021 Jun 10. No abstract available. PMID 34000072